CLINICAL TRIAL: NCT06866782
Title: European Registry of Next Generation Imaging in Advanced Prostate Cancer
Acronym: RING
Status: Recruiting | Type: Observational
Sponsor: Fundacio Puigvert (Other)
Collaborators: European Association of Urology Research Foundation (Other); GUARD Consortium (Genitourinary Alliance for Research and Development) (Unknown); European Association of Urology - Section of Urological Imaging (Unknown); Johnson & Johnson (Industry); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Francesco Sanguedolce, Chief Investigator, Fundacio Puigvert
Other Study IDs: 56021927PCR4037
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Advanced Prostate Cancer; Metastatic Prostate Cancer (mPC)
Keywords: prostate cancer; advanced prostate cancer; new generation imaging; conventional imaging; Metastatic Prostate Cancer; Magnetic Resonance Imaging; PET/CT PSMA; Prostate-Specific Membrane Antigen; Imaging Biomarkers; bone scan; CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- New generation imaging: Patients with prostate cancer at high risk for harbouring metastatic deposits at the hormone-sensitive stage, who require imaging exploration either at the diagnostic workup of a "naïve" patient or at biochemical relapse/progression after local treatment with the use of next generation imaging ( whole-body MRI and PET/CT with new tracers (F/Ga-PSMA, 18F-fluciclovine)
  Interventions: Diagnostic Test: Imaging
- Conventional imaging: Patients with prostate cancer at high risk for harbouring metastatic deposits at the hormone-sensitive stage, who require imaging exploration either at the diagnostic workup of a "naïve" patient or at biochemical relapse/progression after local treatment with the use of conventional imaging ( CT and bone scan)
  Interventions: Diagnostic Test: Imaging
- Conventional imaging and New generation imaging: Patients with prostate cancer at high risk for harbouring metastatic deposits at the hormone-sensitive stage, who require imaging exploration either at the diagnostic workup of a "naïve" patient or at biochemical relapse/progression after local treatment with the use of conventional imaging ( CT and bone scan) AND next generation imaging
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Imaging will be done according to local protocols and/or guidelines of EAU
  Other Names: whole-body MRI; PSMA PET/CT; 18F-fluciclovine PET/CT; Bone Scan; CT; Choline PET/CT

SUMMARY:
The RING study is a European registry collecting real-world data on advanced prostate cancer (APC) imaging. It aims to evaluate the role of next-generation imaging (NGI), such as PET/CT and whole-body MRI, in detecting and monitoring the disease compared to conventional imaging.

Men aged 18 or older with histologically confirmed prostate cancer are eligible to participate in the study if they require imaging to assess potential metastases, either at diagnosis or after relapse and sign a consent form.

Patients will receive standard care with no experimental treatments. Imaging and treatment decisions will follow routine clinical practice. Data will be collected from medical records and analysed for research. This study will help doctors understand when NGI should be used, how it affects treatment decisions, and its impact on patient outcomes.

DETAILED DESCRIPTION:
This registry is intended to collect real-world data on patient demographics, medical history, clinical endpoints, histological tumour characteristics and imaging explorations of the patients with prostate cancer at high risk for harbouring metastatic deposits at the hormone-sensitive stage, who require imaging exploration (conventional, NGI, or their combination) either at the diagnostic workup of a "naïve" patient or at biochemical relapse/progression after local treatment.

Stage 1: cross-sectional observation

1. To identify the proportion of patients for whom an imaging work-up with NGI at baseline may result beneficial, according to physician criteria.
2. Assess management prompted by NGI vs. conventional imaging in usual clinical practice.
3. To identify the proportion of patients for whom conventional imaging is considered informative enough for making a clinical decision, according to physician criteria.
4. Stratification of metastatic prostate cancer patients by the number, volume, and location of deposits, according to the different imaging tools employed.
5. Reclassification of HSPC (M0 vs low vs. high volume) based on NGI respect to CI when both imaging modalities are used. Stage 2: longitudinal observation

1. Evaluation of survival outcomes and their relationship with the imaging pathway undertaken (overall and per subgroup of imaging modality). 2. Identification of prognostic factors related to treatment response and disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients (≥18 years with no upper age limit).
2. Histologically proven prostate cancer.
3. Patients who require imaging exploration (conventional, Next-Generation Imaging (NGI), or their combination) at high risk for harbouring metastatic deposits at the hormone-sensitive stage, either at the diagnostic workout of a "naïve" patient or at biochemical relapse/progression after local treatment.
4. Patients who authorize their participation in the study by signing a written informed consent form (ICF).

Exclusion Criteria:

1. Patients participating in other interventional or non-interventional study which requires NGI as a triage test for metastatic assessment.
2. Patients with evidence of any other clinically significant disease or condition which in the opinion of the investigator discourages their participation in the study.
3. Patients who will not be able to complete the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient "naive" or relapsed/progressed patients above 18 years with prostate cancer at high risk for harbouring metastatic deposits at the hormone-sensitive stage, who require imaging exploration (conventional, NGI, or their combination)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring NGI, conventional imaging, or a combination of both imaging tools. | 4 - 6 weeks
  Number of patients who require NGI, conventional imaging, or a combination of both imaging tools with the respect to local protocols
Proportion of patients with a change of treatment determined by the imaging test result, when multiple imaging tests have been realized | 4-6 weeks
  Number of patients who received multiple imaging tests for whom the result of the particular imaging test has lead to the change in management

OTHER OUTCOMES:
Clinical variables associated to NGI or conventional imaging | 4-6 weeks
  The investigators aim to identify which clinical characteristics (age, ethnicity, comorbidities, PSA, PSA doubling time, ISUP grade at biopsy or at specimens, etc), are associated to the clinical decision of undertaking a systemic work-up with either NGI or CI. This outcome will be measured by means of a univariate and multivariate statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sanguedolce, MD, PhD, Study Chair — Fundació Puigvert
Locations (23):
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- France (3):
  - Hospital Center University De Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - University Hospitals Pitié Salpêtrière, Paris
- Germany (5):
  - Bonn University Hospital, Bonn
  - Martini Klinik, Hamburg
  - München LMU L MU-University Clinic, Munich
  - Urologische Klinik München - Planegg, Planegg
  - Universitätsklinik Tübingen, Tübingen
- Italy (3):
  - IRCCS Universit of Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Ospedale San Raffaele, Milan
- ERASMUS MC & Franciscus Hospital, Rotterdam, Netherlands
- Uniwersytet Jagielloński Collegium Medicum, Krakow, Poland
- Spain (8):
  - Fundació Puigvert, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
- Skånes universitetssjukhus Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
GDPR regulations

REFERENCES:
- [Derived] Chernysheva D, Fanti S, Bjartell A, Afferi L, Breda A, Palou J, Padhani AR, Sanguedolce F. European Registry of Next Generation Imaging in Advanced Prostate Cancer (RING): protocol for an international, prospective registry study. BMJ Open. 2025 Dec 3;15(12):e106022. doi: 10.1136/bmjopen-2025-106022. PMID 41338644

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT06866782/Prot_SAP_000.pdf